CLINICAL TRIAL: NCT06107790
Title: Phase III Clinical Trial Comparing the Safety, Efficacy, and Immunogenicity of HS022 and Trastuzumab® in Combination With Vinorelbine Bitartrate Injection in the Treatment of HER2-positive Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zhejiang Hisun Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HS022-III
Record Dates: First submitted 2023-03-16; First posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-09

CONDITIONS: HER2-positive Breast Cancer
MeSH Terms: interventions — Trastuzumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HS022+ Vinorelbine Bitartrate (Experimental)
  Interventions: Drug: HS022; Drug: Vinorelbine Bitartrate
- Trastuzumab®+ Vinorelbine Bitartrate Injection (Active Comparator)
  Interventions: Drug: Trastuzumab; Drug: Vinorelbine Bitartrate

INTERVENTIONS:
Drug: HS022 — 8 treatment cycles, 3 weeks/cycle, 24 weeks. The first dose is 8 mg/kg , and then 6 mg/kg .3 weeks/cycle, continue until the disease progresses, intolerable toxic reaction occurs, or the subject voluntarily withdraws from the clinical trial, whichever occurs first.
  The second stage 9 treatment cycles, 3 weeks/cycle, 27 weeks. 6mg/kg
  Arms: HS022+ Vinorelbine Bitartrate
Drug: Trastuzumab — 8 treatment cycles, 3 weeks/cycle, 24 weeks. The first dose is 8 mg/kg , and then 6 mg/kg .3 weeks/cycle, continue until the disease progresses, intolerable toxic reaction occurs, or the subject voluntarily withdraws from the clinical trial, whichever occurs first.
  The second stage 9 treatment cycles, 3 weeks/cycle, 27 weeks. 6mg/kg
  Arms: Trastuzumab®+ Vinorelbine Bitartrate Injection
Drug: Vinorelbine Bitartrate — Vinorelbine: 25mg/m2 (intravenous infusion, day 1 and 8 of each cycle). 3 weeks/cycle, continue until the disease progresses, intolerable toxic reaction occurs, or the subject voluntarily withdraws from the clinical trial, whichever occurs first.
  Second section:9 treatment cycles, 3 weeks/cycle, 27 weeks. Vinorelbine: 25mg/m2 (intravenous infusion, day 1 and 8 of each cycle). The investigator may decide whether to continue treatment with vinorelbine at his discretion.
  3 weeks/cycle, continue until the disease progresses, intolerable toxic reaction occurs, or the subject voluntarily withdraws from the clinical trial, whichever occurs first.

SUMMARY:
This is a multi-center, randomized, double-blind, parallel-group study to evaluate the efficacy and safety and Immunogenicity of Vinorelbine Bitartrate Injection in Combination With HS022 and Trastuzumab®.There were 2 parts. Part 1 needs 8 treatment cycles ( at least 24 weeks); Part2 needs 9 treatment cycles (at least 27 weeks).

ELIGIBILITY:
Inclusion Criteria:

* 1. Female ≥18 and ≤75 years of age on day of signing the informed consent form (ICF).

  2. Histologically or cytologically confirmed adenocarcinoma of the breast. 3. Recurrent disease not amenable to curative surgery or radiation therapy. 4. HER2-positivity, based on IHC score 3+ or ISH positivity. For those IHC score 2+ patients, fluorescence in situ hybridization (FISH), chromogenic in situ hybridization (CISH) or silver enhanced in situ hybridization (SISH) should be tested to prove HER2 gene amplification.

  5.No prior systemic anticancer agent such as chemotherapy, biological or targeted agent for metastatic disease. For patients with recurrent disease, prior neo-/adjuvant therapy containing trastuzumab must have been stopped at least 12 months before the diagnosis of recurrent (local or metastatic) disease.

  6.Those with at least one measurable target lesion (RECIST 1.1 standard): at least one diameter line of the target lesion can be accurately measured, and the lesions, skin lesions, brain lesions, and bone metastases of any type after radiotherapy or other local regional treatment can only be evaluated as non-target lesions; 7.ECOG < 2； 8.Left ventricular ejection fraction (LVEF) ≥ 50% within 4 weeks before randomization; 9.Adequate hematology, liver function and kidney function, as shown in the following laboratory test values；

  .a) Absolute value of neutrophil ≥ 1.5 × 109/L； b) Platelet ≥ 100 × 109/L, and hemoglobin ≥ 90g/L; c) Total serum bilirubin ≤ 1.5 times the upper limit of normal value (except for Gilbert syndrome); d) ALT and AST ≤ 2.5 times the upper limit of normal value (subjects with liver metastasis ≤ 5 times the upper limit of normal value); e) Blood creatinine ≤ 1.5 times the upper limit of normal value. 10.The expected survival period ≥ 3 months. 11. Patients have voluntarily agreed to participate and given written informed consent.

Exclusion Criteria:

* .Prior surgery within 4 weeks preceeding enrollment or expected to be performed during the trial, prior chemotherapy wihtin 4 weeks preceeding enrollment, prior radiotherapy or endocrinotherapy within 4 weeks before enrollment.

  2.Prior treatment with vinorelbine 3.Current peripheral neuropathy above 2 grades 4.Known brain metastasis or other CNS metastasis that is either symptomatic or untreated. Central nervous system metastases that have been treated by complete resection and/or radiotherapy demonstrating stability or improvement are not an exclusion criterion provided they are stable as shown by computed tomography (CT) or magnetic resonance imaging (MRI) scan for at least 4 weeks before Screening without evidence of cerebral edema and no requirements for corticosteroids or anticonvulsants.

  5.Participation in another clinical study within 4 weeks before enrollment (3 months for studies involving monoclonal therapy), excluding those who failed in screening;

  6. Patients with any other malignant tumor in the past five years, excluding fully cured cervical carcinoma in situ, basal cell or squamous cell skin cancer;

  7. Have a clear history of neurological or mental disorders, including epilepsy or dementia;

  8. Those who are allergic to any ingredient or excipient of the test drug, including those who are allergic to benzyl alcohol;

  9. Those who have received whole blood or component blood transfusion within 2 weeks before randomization;

  10. Those who currently suffer from diseases affecting intravenous injection and venous blood collection;

  11. At present, there are serious and uncontrollable systemic diseases (such as dyspnea, bronchospasm, acute attack of asthma or other diseases requiring continuous oxygen inhalation treatment), which, according to the judgment of the researcher, will significantly affect the participation/completion of the test and efficacy evaluation of the subjects;

  12. Have any of the following heart diseases:
  1. Currently suffering from untreated or uncontrollable hypertension (systolic blood pressure>150 mmHg or diastolic blood pressure>100 mmHg), or unstable angina pectoris;
  2. According to the standards of the New York Heart Association, he currently has a history of congestive heart failure at any level, or serious arrhythmia requiring treatment (excluding atrial fibrillation or paroxysmal supraventricular tachycardia);
  3. Myocardial infarction occurred within 6 months before signing the informed consent;

     13. At present, people who need to use corticosteroids daily for long-term treatment (the equivalent dose of methylprednisolone with dose>10 mg/day), excluding inhaled corticosteroids; 14. Any one of human immunodeficiency virus antibody, treponema pallidum antibody and hepatitis C virus antibody should be excluded. Or there are patients with active hepatitis B infection of clinical significance who need treatment: hepatitis B surface antigen [HBsAg] or hepatitis B core antibody [HBcAb] is positive, and hepatitis B virus deoxyribonucleic acid [HBV DNA] test results are greater than or equal to the upper limit of the reference value of each hospital. Among them, only those with positive syphilis specific antibody test but negative syphilis non-specific antibody test can be selected; Only those with positive hepatitis C virus antibody but negative hepatitis C virus RNA [HCV RNA] can be selected;;

     15. Pregnant or lactating women; Or when screening, the blood pregnancy test of women of childbearing age is positive; Or women of childbearing age and their spouses are unwilling to take effective contraceptive measures during and within 7 months after the end of the clinical trial;

     The researcher believes that it is not suitable for enrollment or may not be able to complete the test for other reasons.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 570 (Actual)
Dates: Start 2018-05-16 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2022-01-28 (Actual)

PRIMARY OUTCOMES:
ORR | WEEK 25
  The best overall response rate (ORR24: performed at the 25th week): According to the Solid Tumor Efficacy Evaluation Standard (RECIST) 1.1, the proportion of CR and PR subjects from the first evaluation (baseline) to the 25th week of treatment (after the completion of 8 treatment cycles) (note: including unconfirmed response).

SECONDARY OUTCOMES:
DCR | WEEK 25
  Disease control rate (DCR: in the 25th week): DCR=CR+PR+SD。
PFS | WEEK 52
  Progression-free survival (PFS: the 52nd week): according to RECIST1.1, the time from the date of randomization to the date of disease progression or all-cause death (whichever occurs first). If the subjects did not have the above events, the PFS would be closed to the date of the last full tumor evaluation.
OS | WEEK 52
  Total survival rate (OS rate: performed at the 52nd week): defined as the percentage of subjects who survived at 51 weeks after randomization.
Vital signs | first day and the 8th day at each visit prior to administration（1st cycle , the 2nd cycle, the 3rd cycle, the 4th cycle the 5th cycle, the 6th cycle,the 7th cycle,the 8th cycle,or the 22nd day after the last administration of the early withdrawal.
  temprature
Vital signs | first day and the 8th day at each visit prior to administration（1st cycle , the 2nd cycle, the 3rd cycle, the 4th cycle the 5th cycle, the 6th cycle,the 7th cycle,the 8th cycle,or the 22nd day after the last administration of the early withdrawal.
  pulse rate
Vital signs | first day and the 8th day at each visit prior to administration（1st cycle , the 2nd cycle, the 3rd cycle, the 4th cycle the 5th cycle, the 6th cycle,the 7th cycle,the 8th cycle,or the 22nd day after the last administration of the early withdrawal.
  respiration（in times/minute）
Vital signs | first day and the 8th day at each visit prior to administration（1st cycle , the 2nd cycle, the 3rd cycle, the 4th cycle the 5th cycle, the 6th cycle,the 7th cycle,the 8th cycle,or the 22nd day after the last administration of the early withdrawal.
  blood pressure (systolic/diastolic，in mmHg)
physical examination, | first day and the 8th day at each visit prior to administration（1st cycle , the 2nd cycle, the 3rd cycle, the 4th cycle the 5th cycle, the 6th cycle,the 7th cycle,the 8th cycle,or the 22nd day after the last administration of the early withdrawal.
  Perform a physical examination at each visit
ADAs | on the 22nd day after the last administration
  The incidence of anti-drug antibodies (ADAs) before treatment, after 2 cycles of treatment, after 4 cycles, after 6 cycles, after 8 cycles, after 12 cycles, on the 22nd day after the last administration of 17 cycles/on the 22nd day after the last administration (test/non test drug) of early withdrawal
Ctrough | In two hours before the administration of the trial drug on the first day of the 1st, 3rd, 5th and 7th cycles, the 22nd day of the 8th cycle)/the 22nd day after the last administration. Each cycle was 21 days.
  Collect serum samples for PK testing according to the protocol/laboratory manual, and transport them to the biological sample analysis laboratory for unified testing and analysis
ECOG physical condition | first day and the 8th day at each visit prior to administration（1st cycle , the 2nd cycle, the 3rd cycle, the 4th cycle the 5th cycle, the 6th cycle,the 7th cycle,the 8th cycle,or the 22nd day after the last administration of the early withdrawal.
  ECOG physical condition
left ventricular ejection fraction (LVEF), | first day and the 8th day at each visit prior to administration（1st cycle , the 2nd cycle, the 3rd cycle, the 4th cycle the 5th cycle, the 6th cycle,the 7th cycle,the 8th cycle,or the 22nd day after the last administration of the early withdrawal.
  left ventricular ejection fraction (LVEF),
adverse events (AE) | first day and the 8th day at each visit prior to administration（1st cycle , the 2nd cycle, the 3rd cycle, the 4th cycle the 5th cycle, the 6th cycle,the 7th cycle,the 8th cycle,or the 22nd day after the last administration of the early withdrawal.
  adverse events (AE)

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Province People's Hospital (First Affiliated Hospital of Nanjing Medical University), Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided